CLINICAL TRIAL: NCT01099813
Title: The Effect of Pathophysiological and Organisational Lead Times to Critical Care on Survival and Resource Utilisation
Brief Title: Sepsis Pathophysiological & Organisational Timing
Acronym: SPOT(Light)
Status: Completed | Type: Observational
Sponsor: Intensive Care National Audit & Research Centre (Other)
Collaborators: Wellcome Trust (Other); London School of Hygiene and Tropical Medicine (Other)
Responsible Party: Principal Investigator, Steve Harris, Dr, University College, London
Other Study IDs: SPOT-Light
Record Dates: First submitted 2010-04-07; First posted 2010-04-08 (Estimated); Last update posted 2014-05-23 (Estimated); Status verified 2014-05

CONDITIONS: Critical Illness; Sepsis
Keywords: Critical Illness; Sepsis; Duration; Severity of Illness Scores; Trajectory
MeSH Terms: conditions — Critical Illness; Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Inpatients assessed for critical care: Patients admitted to Critical Care Units participating in the ICNARC CMP programme who have been assessed at any time on a ward prior to ICU admission by a critical care decision maker (e.g. the CCOT or any member of the medical staff on duty for the unit)

SUMMARY:
This project proposes to measure delay to admission to Intensive Care (ICU). Delays in the United Kingdom NHS are widely reported possibly because there are fewer ICU beds than in many other developed health care systems. Patients are inevitably admitted with more severe illness. Scores measuring this severity are used for research and benchmarking. However, although patients deteriorate over time, severity is probably neither directly nor linearly related to the duration of illness. Instead it is likely that the characteristics of severity change with time. In sepsis there is good biological evidence of this so that there is an early pro-inflammatory stage followed by later changes in metabolic, neuroendocrine, and immune systems. In addition to examining the effect of duration of illness prior to ICU admission, the investigators will also therefore investigate how severity changes over time.

SPOT(Light) is a prospective observational study. Treatment is not modified in anyway. Patients evaluated on the ward by critical care outreach teams, and subsequently admitted to critical care will be eligible. Severity of illness at the time of initial evaluation and eventual admission will be compared, and the effect of the duration of illness on 90 day survival investigated.

DETAILED DESCRIPTION:
It is useful to consider time in critical illness from two perspectives. The first of these begins logically with onset of the pathology. With the exception of conditions such as myocardial infarction or trauma where this moment is marked by a classic symptom or an external event, then defining time zero is difficult. For this reason, an organisational frame of reference, such as hospital admission or time of referral to specialist team, is more commonly used. Delay following this organisational time is important because it is often a modifiable factor with regard to the delivery of health care. However, pathophysiological timing remains relevant because if the disease process is dynamic (and this is part of the hypothesis of this study) then it determines the phenotype of disease at any particular moment.

This project proposes to measure delay to admission to Intensive Care (ICU) using both organisational and pathophysiological timing. Delays in the United Kingdom NHS are widely reported {McQuillan:1998p127, Hillman:2001p90} possibly because there are fewer ICU beds than in many other developed health care systems.{Wunsch:2008p121} We intend to measure the chronological time between the moment when a patient is 'referred and assessed as requiring Critical Care', and their actual time of admission. We will determine how often delays occur, and whether they affect outcome. Requirements for critical care are not, however, absolute. Importantly, the assessment of a prospective patient is not made in isolation. If ICU beds are already fully occupied, then decision makers must organise a transfer to another unit (with risks to the patient), organise a premature discharge of another patient, or defer admission. We will also therefore consider such deferments alongside delays, and their impact on survival.

In addition, the project will consider pathophysiological timing. This is of particular importance in sepsis where current biological models suggest that there is a phased response to infection.{Riedemann:2003p82} In this case, it is possible that patients are admitted to critical care at different phases of disease; moreover, these phases may be clinically relevant and affect response to treatment. pathophysiological delay will be estimated using the concept of illness trajectories (which also may have a biological correlate){Osuchowski:2006p2107}. This means that a patient who is slowly deteriorating is likely to have been ill for longer. In other words, their pathophysiological time zero will be earlier than another patient who is is rapidly deteriorating. This illness trajectory will be estimated by measuring the change in severity of illness between ward assessment and ICU admission. The effect of these illness trajectories, and therefore of the pathophysiological timing of ICU admission, will be evaluated with particular attention to severe sepsis.

ELIGIBILITY:
Exclusion Criteria:

* Paediatric patients (Age < 18 years)
* Elective or planned admissions to critical care

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to Critical Care Units participating in the ICNARC CMP programme who have been assessed at any time on a ward prior to ICU admission by a critical care decision maker (e.g. the CCOT or any member of the medical staff on duty for the unit)
Sampling Method: Non-Probability Sample
Enrollment: 15602 (Actual)
Dates: Start 2010-11; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Survival | 90 day

CONTACTS AND LOCATIONS:
Overall Officials: Steve Harris, MRCP FRCA, Principal Investigator — ICNARC / LSHTM
Locations (1):
- University College Hospital London, London, London, United Kingdom

REFERENCES:
- See also: Intensive Care National Audit & Research Centre — https://www.icnarc.org/Our-Research/Studies/Spotlight/About